CLINICAL TRIAL: NCT05060120
Title: Biomarker Panel for Early Diagnosis of Ovarian Torsion
Brief Title: Biomarker Panel in Ovarian Torsion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Principal Investigator, Oshri Barell, head of gynecology unit, Assuta Ashdod Hospital
Other Study IDs: AAA-21-0094
Record Dates: First submitted 2021-09-12; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Ovary Torsion; Adnexal Torsion
MeSH Terms: conditions — Ovarian Torsion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and peritoneal fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- confirmed ovarian torsion: immediately before laparoscopy and 1 day post- operation and four weeks after laparoscopy a panel of serum biomarkers will be tested
  Interventions: Diagnostic Test: biomakers for ovarian torsion; Diagnostic Test: peritoneal fluid proteins analysis
- confirmed non ovarian torsion: immediately before laparoscopy
  Interventions: Diagnostic Test: biomakers for ovarian torsion
- control group: match control Compare healthy controls with patients with or without ovarian torsion as confirmed by laparoscopy
  Interventions: Diagnostic Test: biomakers for ovarian torsion

INTERVENTIONS:
Diagnostic Test: biomakers for ovarian torsion — Blood biomarkers analysis using multiplex ELISA: The Luminex system is a magnetic bead-based multiplex ELISA that enable to measure simultaneously multiple proteins within the same sample. Human magnetic Luminex assay will be used for the following analytes: D-Dimer (21.7-5,280 ng/ml), FABP4/A-FABP (0.637-155 ng/ml), GM-CSF (0.012-2.98 ng/ml), ICAM-1/CD54 (6.9-1674 ng/ml), IFN-γ (0.058-14.2 ng/ml), IL-1α (0.005-1.27 ng/ml), IL-6 (0.005-1.2 ng/ml), IL-10 (0.005-1.2 ng/ml), IL-17/IL-17A (0.012-3.1 ng/ml), Park7/DJ-1 (0.26- 63.1 ng/ml), TNF-α (0.01-2.4 ng/ml), TSLP (0.003-0.7 ng/ml), VCAM-1/CD106 (7.8-1891 ng/ml) and VEGF (0.008-2.4 ng/ml). Plasma samples stored at -70°C will be sent to accredited lab at BioTest (Israel) for performing the multiplex ELISA readout assay test using MagPix system.
Diagnostic Test: peritoneal fluid proteins analysis — Western blot for peritoneal fluid proteins analysis
  We will look for the relative abundance of proteins involved in the protection of cells against oxidative stress and the regulation of reactive oxygen species (ROS) using western blot. Superoxide dismutase 1 (SOD1, 16kDa) scavenges superoxides (O-2) within cells. Catalase (60kDa) is hydrogen peroxide (H2O2) scavenging enzyme regulate ROS concentrations within cells by reducing H202 into O2 and water. Thioredoxin (12kDa) facilitates the reduction of proteins via cysteine thiol-disulfide exchange. Alpha smooth muscle actin (42kDa) will be used as a loading control. These four proteins will be resolved by western blot given their different molecular weights using western blot cocktail antibodies (abcam # ab179843).
  Groups: confirmed ovarian torsion

SUMMARY:
The overall goal of the project is to find a panel of novel biomarkers for early detection of ovarian torsion.

DETAILED DESCRIPTION:
The overall goal of the project is to find a panel of novel biomarkers for early detection of ovarian torsion.

The specifc aims of the current study are:

1. Screen for changes in blood protein biomarkers concentrations specifc for patients with ovarian torsion. The biomarkers are: D-Dimer (21.7-5,280 ng/ml), FABP4/A-FABP (0.637-155 ng/ml), GM-CSF (0.012-2.98 ng/ml), ICAM-1/CD54 (6.9-1674 ng/ml), IFN-γ (0.058-14.2 ng/ml), IL-1α (0.005-1.27 ng/ml), IL-6 (0.005-1.2 ng/ml), IL-10 (0.005-1.2 ng/ml), IL-17/IL-17A (0.012-3.1 ng/ml), Park7/DJ-1 (0.26- 63.1 ng/ml), TNF-α (0.01-2.4 ng/ml), TSLP (0.003-0.7 ng/ml), VCAM-1/CD106 (7.8-1891 ng/ml) and VEGF (0.008-2.4 ng/ml).
2. Compare the amount of oxidative stress defense proteins SOD1, Catalase, and Thioredoxin amount in the peritoneal fluid wash between patients with or without confirmed ovarian torsion. To our knowledge, this is the first study that specifically evaluates the expression of oxidation stress defense proteins in ovarian torsion. The results will enable us to decide whether to include oxidation stress biomarkers within the panel.
3. Study population methodology and techniques

A prospective, 12-24 months study.

20 Patients with confirmed ovarian torsion will be enrolled.

The patients will complete a questionnaire prior to and following the procedure

3.5ml blood samples will be obtained immediately before laparoscopy, postoperative day, and four weeks after laparoscopy during the follow-up.

The peritoneal fluid wash will be collected during the laparoscopy from 14 patients (out of the 20 enrolled) that will provide additional written consent specific for the procedure.

20 Patients suspected of ovarian torsion with no ovarian torsion, as confirmed by laparoscopy, will be enrolled.

The patients will complete a questionnaire prior to and following the procedure

5ml blood samples will be obtained immediately before laparoscopy and four weeks after laparoscopy during the follow-up.

The peritoneal fluid wash will be collected during the laparoscopy from 14 patients (out of the 20 enrolled) that will provide additional written consent specific for the procedure.

20 Healthy controls will be enrolled and provide a 5ml blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 12 and 50 years who were admitted to the gynecological emergency room at Assuta medical center with signs and symptoms suggestive of ovarian torsion
* Patients that will undergo laparoscopy for the diagnosis of ovarian torsion
* Able to provide informed consent for themselves or have a legal guardian that can provide informed consent (in cases of patients under 18 years old)

Exclusion criteria:

* Patients that are unable to provide informed consent

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Female patients between 12 and 50 years, who were admitted to the gynecological emergency room at Assuta medical center with signs and symptoms suggestive of ovarian torsion.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
preoperative biochemical test -BIOMARKER PANEL FOR OVARIAN TORSION | 2 years
  Screen for elevation in blood protein biomarkers concentrations specifc for patients with ovarian torsion. The biomarkers are: D-Dimer (21.7-5,280 ng/ml), FABP4/A-FABP (0.637-155 ng/ml), GM-CSF (0.012-2.98 ng/ml), ICAM-1/CD54 (6.9-1674 ng/ml), IFN-γ (0.058-14.2 ng/ml), IL-1α (0.005-1.27 ng/ml), IL-6 (0.005-1.2 ng/ml), IL-10 (0.005-1.2 ng/ml), IL-17/IL-17A (0.012-3.1 ng/ml), Park7/DJ-1 (0.26- 63.1 ng/ml), TNF-α (0.01-2.4 ng/ml), TSLP (0.003-0.7 ng/ml), VCAM-1/CD106 (7.8-1891 ng/ml) and VEGF (0.008-2.4 ng/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Batel Hamou, MD, Principal Investigator — Assuta Ashdod University Hospital
Locations (1):
- Assuta Ashdod University Hospital, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swenson DW, Lourenco AP, Beaudoin FL, Grand DJ, Killelea AG, McGregor AJ. Ovarian torsion: Case-control study comparing the sensitivity and specificity of ultrasonography and computed tomography for diagnosis in the emergency department. Eur J Radiol. 2014 Apr;83(4):733-8. doi: 10.1016/j.ejrad.2014.01.001. Epub 2014 Jan 8. PMID 24480106
- [Background] Cohen SB, Wattiez A, Stockheim D, Seidman DS, Lidor AL, Mashiach S, Goldenberg M. The accuracy of serum interleukin-6 and tumour necrosis factor as markers for ovarian torsion. Hum Reprod. 2001 Oct;16(10):2195-7. doi: 10.1093/humrep/16.10.2195. PMID 11574515
- [Background] Boaz M, Chernin G, Schwartz I, Katzir Z, Schwartz D, Agbaria A, Gal-Oz A, Weinstein T. C-reactive protein and carotid and femoral intima media thickness: predicting inflammation. Clin Nephrol. 2013 Dec;80(6):449-55. doi: 10.5414/CN108067. PMID 24131677
- [Background] Kart C, Aran T, Guven S, Karahan SC, Yulug E. Acute increase in plasma D-dimer level in ovarian torsion: an experimental study. Hum Reprod. 2011 Mar;26(3):564-8. doi: 10.1093/humrep/deq378. Epub 2011 Jan 17. PMID 21242148
- [Background] Guven S, Kart C, Guvendag Guven ES, Cetin EC, Mentese A. Is the measurement of serum ischemia-modified albumin the best test to diagnose ovarian torsion? Gynecol Obstet Invest. 2015;79(4):269-75. doi: 10.1159/000367787. Epub 2015 Jan 9. PMID 25591981
- [Background] Khreiss T, Jozsef L, Potempa LA, Filep JG. Conformational rearrangement in C-reactive protein is required for proinflammatory actions on human endothelial cells. Circulation. 2004 Apr 27;109(16):2016-22. doi: 10.1161/01.CIR.0000125527.41598.68. Epub 2004 Mar 29. PMID 15051635
- [Background] Uyanikoglu H, Hilali NG, Yardimciel M, Koyuncu I. A new biomarker for the early diagnosis of ovarian torsion: SCUBE-1. Clin Exp Reprod Med. 2018 Jun;45(2):94-99. doi: 10.5653/cerm.2018.45.2.94. Epub 2018 Jun 29. PMID 29984210
- [Result] Piper HG, Oltmann SC, Xu L, Adusumilli S, Fischer AC. Ovarian torsion: diagnosis of inclusion mandates earlier intervention. J Pediatr Surg. 2012 Nov;47(11):2071-6. doi: 10.1016/j.jpedsurg.2012.06.011. PMID 23164000